CLINICAL TRIAL: NCT01824979
Title: Pilairo Lab Market Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIA76
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Results first posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pilairo mask (Experimental): Pilairo nasal pillows mask during CPAP titration
  Interventions: Device: CPAP mask ( Pilairo)
- Other CPAP mask (Active Comparator): Other CPAP mask during CPAP titration
  Interventions: Procedure: Other CPAP mask

INTERVENTIONS:
Device: CPAP mask ( Pilairo)
  Arms: Pilairo mask
Procedure: Other CPAP mask
  Arms: Other CPAP mask

SUMMARY:
The purpose of the study is to observe the Pilairo mask in a lab setting.

DETAILED DESCRIPTION:
The purpose of the study is to observe the Pilairo mask in a lab setting, compared to other commercially available masks for continuous positive airwary pressure (CPAP) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Apnea Hypopnea Indea >15 from diagnostic study
* Minimum 18 years of age

Exclusion Criteria:

* Inability ot give informed consent
* History of intolerance to CPAP
* Anatomical or physiological conditions making CPAP therapy inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Peninsula Sleep Center Inc, Burlingame, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilairo: Pilairo nasal pillows mask during CPAP titration
  CPAP mask ( Pilairo)
- Other CPAP Mask: Other CPAP mask during CPAP titration
  Other CPAP mask
Period: Overall Study
Arm/Group | Pilairo | Other CPAP Mask
Started | 50 | 50
Completed | 37 | 37
Not Completed | 13 | 13
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilairo | Other CPAP Mask | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Count of Participants; unit: Participants] — Inclusion criteria only confirmed participants were over the age of 18. Full date of birth was not recorded on the case report form. Therefore, the exact breakdown of participants in each age bracket is unable to be provided as is required in the non-customized Baseline measure.
  Participants
    ≥ 18 years | 50 | 50 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 19 | 29
  Male | 40 | 31 | 71
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Technician Experience With Mask
Description: Measured from a single item, sleep technicians indicated their experience using the Pilairo or Other CPAP mask during the CPAP titration. Response options ranged on a scale from 0 to 10 with 0 indicating an extremely poor experience and 10 indicating and extremely pleasant experience.
Time Frame: One night
Population: While not all participants completed the full study, a number of participants had completed enough of the study to provide data to analyze. For this outcome measure, 48 participants in the Pilairo Group had usable data for analysis while 42 participants in the Other CPAP mask group had usable data for analysis for this measure.
Measure: Mean (Full Range); unit: Units on a Scale
Arm/Group | Pilairo | Other CPAP Mask
Number analyzed (Participants) | 48 | 42
Units on a Scale | 8.46 [0 to 10] | 8.24 [0 to 10]

2. Secondary Outcome: Number of Mask Interventions During the Night
Description: Sleep technicians reported the number of times they had to intervene with the mask to get a good seal or improve comfort.
Time Frame: One night
Population: as for outcome 1
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Pilairo | Other CPAP Mask
Number analyzed (Participants) | 48 | 42
units on a scale | 1.29 [0 to 5] | 2.20 [0 to 5]

ADVERSE EVENTS:
Time Frame: 1 night in lab
Arm/Group | Pilairo | Other CPAP Mask
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No